CLINICAL TRIAL: NCT00803725
Title: Spinal Mepivicaine With Fentanyl for Outpatient Knee Arthroscopy Surgery
Brief Title: Spinal Mepivicaine With Fentanyl for Outpatient Knee Arthroscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Dr. Richard Brull, University Health Network
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 07-0683-A
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Last update posted 2010-01-26 (Estimated); Status verified 2010-01

CONDITIONS: Knee Arthroscopy
Keywords: spinal anesthesia; mepivacaine; fentanyl; duration of anesthesia; knee arthroscopy; regional anesthesia; Spinal anesthesia for knee arthroscopy
MeSH Terms: interventions — Mepivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Mepivicaine for spinal anesthesia
  Interventions: Drug: Mepivacaine without fentanyl
- 2 (Experimental): Mepivacaine with Fentanyl for spinal anesthesia
  Interventions: Drug: Mepivacaine with Fentanyl

INTERVENTIONS:
Drug: Mepivacaine without fentanyl — 45 mg 1.5% mepivacaine injection for spinal anesthesia
  Arms: 1
Drug: Mepivacaine with Fentanyl — 10 micrograms fentanyl with 30 mg 1.5% mepivacaine injection for spinal anesthesia
  Arms: 2

SUMMARY:
The purpose of this study is to determine if the addition of intrathecal fentanyl to low dose mepivacaine spinal anesthesia provides adequate surgical anesthesia with shorter duration of motor blockade.

It is hypothesized that lower doses of spinal mepivacaine when combined with fentanyl will result in adequate surgical block for knee arthroscopy surgery with faster recovery and discharge compared to mepivacaine alone.

ELIGIBILITY:
Inclusion Criteria:

1. Patients having unilateral arthroscopic surgery of the knee;
2. ASA I-III status;
3. Age 18-80 years;
4. BMI< 35.

Exclusion Criteria:

1. Patients who have previous history of hypersensitivity to local anesthetics or contraindications for spinal anesthesia (i.e. bleeding diathesis, coagulopathy);
2. Patients with radiating low back pain and neurological deficits in lower extremities;
3. Patients who are incapable of giving an informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Time to complete motor block regression (0) as measured by modified Bromage scale. | Every 2 minutes from administration of the spinal until complete onset.

SECONDARY OUTCOMES:
Block success, peak, and duration; time to ambulation, urination, discharge; incidence of adverse events. | Up to 72 hours after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] O'Donnell D, Manickam B, Perlas A, Karkhanis R, Chan VW, Syed K, Brull R. Spinal mepivacaine with fentanyl for outpatient knee arthroscopy surgery: a randomized controlled trial. Can J Anaesth. 2010 Jan;57(1):32-8. doi: 10.1007/s12630-009-9207-6. Epub 2009 Oct 24. PMID 19856040